CLINICAL TRIAL: NCT04152837
Title: An Open-Label Study of Lixivaptan in Subjects With Autosomal Dominant Polycystic Kidney Disease Who Previously Experienced Abnormal Liver Chemistry Test Results While Receiving Tolvaptan: The ALERT Study
Brief Title: Safety of Lixivaptan in Subjects Previously Treated With Tolvaptan for Autosomal Dominant Polycystic Kidney Disease
Acronym: ALERT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The decision is based on a thorough reassessment of the commercial potential of lixivaptan as a potential best-in-class therapy for patients with ADPKD
Sponsor: Palladio Biosciences (Industry)
Collaborators: Centessa Pharmaceuticals plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA-ADPKD-303
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Results first posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Polycystic Kidney Disease, Adult; ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — lixivaptan

STUDY DESIGN:
Intervention Model Description: Open-label, single treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lixivaptan (Experimental): Lixivaptan oral capsules, 100-200 mg twice daily
  Interventions: Drug: Lixivaptan

INTERVENTIONS:
Drug: Lixivaptan — Oral vasopressin V2 receptor antagonist

SUMMARY:
This is a Phase 3, open-label, repeat-dose study designed to assess liver safety, non-liver safety, and efficacy of lixivaptan in participants who previously experienced liver chemistry test abnormalities while treated with tolvaptan and were permanently discontinued from the drug for that reason. Up to 50 eligible participants will be enrolled and treated with lixivaptan for 52 weeks following titration to an optimal dose.

DETAILED DESCRIPTION:
This is a Phase 3, open-label, repeat-dose study designed to assess liver safety, non-liver safety, and efficacy of lixivaptan in participants who previously experienced liver chemistry test abnormalities while treated with tolvaptan and were permanently discontinued from the drug for that reason. Up to 50 participants will be enrolled and treated. Evaluations will include frequent testing of liver chemistry (every week during the Baseline and Titration Periods and every 4 weeks during the Maintenance Period), physical examinations, vital signs, safety labs (serum chemistry, hematology, urinalysis), estimated glomerular filtration rate (eGFR), urine specific gravity and osmolality determinations and trough serum concentration of lixivaptan. After meeting entry criteria during a 1- to 3-week Screening Period that can extend up to 8 weeks for medication adjustment, participants will enter a 3-week no study treatment Baseline Period to obtain baseline measurements followed by a 3- to 6-week Titration Period during which lixivaptan administered twice daily (BID) will be titrated to a dose that is tolerated and results in a reduced trough urine specific gravity, or to the maximum dose level. The minimum dose to enter the Maintenance Period is 100 mg BID. Treatment will continue for up to 52 weeks (12 months) after which study drug will be held, and final assessments obtained during the Follow-up Period of 4 weeks. The total study duration will be up to approximately 73 weeks (16.8 months).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 and 65 years of age (inclusive) at the time of Screening.
* Documented diagnosis of ADPKD by imaging or genetic analysis previously treated with tolvaptan for that indication.
* Screening eGFR ≥ 20 mL/min/1.73 m^2.
* Body mass index (BMI) between 18 and 35 kg/m^2 (inclusive) at the time of Screening.
* Documented history of:

  * Based on upper limit of normal (ULN): At least 2 elevated alanine aminotransferase (ALT) levels; 1 ALT level >2 x ULN and 1 ALT level >3 x ULN while the participant was receiving tolvaptan, or within 4 weeks after tolvaptan discontinuation, with no other explanation for the ALT elevations. The 2 elevated ALT measurements could be recorded during the same instance of liver injury or during distinct instances; OR
  * Based on the participant's stable baseline as determined by the Investigator: At least 2 elevated ALT levels; 1 ALT level >2 x the participant's stable baseline level and 1 ALT level >3 x the participant's stable baseline level while the participant was receiving tolvaptan, or within 4 weeks after tolvaptan discontinuation, with no other explanation for the ALT elevations; provided that at least one ALT elevation was >2 x ULN. The 2 elevated ALT measurements could be recorded during the same instance of liver injury or during distinct instances; OR
  * A pattern of ALT elevations deemed by the Investigator to be consistent with tolvaptan liver injury with no other explanation for the ALT elevations and agreement of the medical monitor and sponsor.
* Permanent discontinuation of prior tolvaptan treatment because of the ALT abnormality.
* If re-challenge with tolvaptan was performed, the ALT level must have increased to >2 x ULN upon rechallenge or the ALT level was increasing but tolvaptan was stopped for patient safety reasons before it reached > 2 x ULN after having previously normalized.
* Appropriate control of hypertension including an angiotensin converting enzyme inhibitor or angiotensin receptor blocker (unless not considered appropriate for the participant) without the use of a diuretic in concert with Kidney Disease: Improving Global Outcomes "Clinical Practice Guideline for the Management of Blood Pressure in Chronic Kidney Disease".

  * Willing to practice acceptable methods of birth control (both males who have partners of child-bearing potential and females of childbearing potential).
  * Able to provide informed consent.

Exclusion Criteria:

* Known sensitivity or idiosyncratic reaction to any compound present in lixivaptan and related compounds.
* Hypovolemia at Screening.
* Abnormal serum sodium concentration at Screening.
* Subjects who have taken any investigational drug or used an investigational device within 30 days, or 5 half-lives, whichever is longer, prior to Screening.
* Subjects who are taking, have taken within the past 2 weeks, or are expected to be taking, strong or moderate CYP3A4 or CYP2C8 inhibitors or inducers including regular use of grapefruit juice, Seville oranges, or St. John's wort.
* Simvastatin at total daily doses >10 mg or amlodipine at total daily doses >5 mg.
* Use of tolvaptan within the 3 months prior to Screening or until a previously elevated ALT level has returned to ≤1 x ULN for at least 3 months.
* Use of lixivaptan or participation in a clinical study with lixivaptan within the 3 months prior to Screening.
* Use of conivaptan, somatostatin analogs (e.g., lanreotide, pasireotide, octreotide, etc.), metformin, nicotinamide, bardoxolone, venglustat, demeclocycline, or mammalian Target of Rapamycin (mTOR) kinase inhibitors (e.g., everolimus, sirolimus, etc.) to treat ADPKD within the 3 months prior to Screening.
* Requirement for chronic diuretic use.
* History of advanced diabetes (e.g., glycosylated hemoglobin [HgbA1c] >7.5%, and/or glycosuria by dipstick, significant proteinuria [>300 mcg albumin/mg creatinine]), other significant renal disease, transplanted kidney, recent kidney surgery within the 6 months prior to Screening (including cyst drainage or fenestration) or acute kidney injury within the 6 months prior to Screening.
* Clinically significant incontinence, overactive bladder, or urinary retention (e.g., benign prostatic hyperplasia).
* New York Heart Association Functional Class 3 or 4 heart failure or other significant cardiac or electrocardiogram (ECG) findings that could pose a safety risk to the participant.
* Clinically significant liver disease or impairment or active chronic hepatitis at Screening.
* Positive test results for hepatitis B surface antigen (HBsAg) or hepatitis C (HCV) antibody.
* History of infection with human immunodeficiency virus (HIV) unless the participant is stable and doing well on a non-CYP interacting anti-retroviral therapy (ART) regimen and who has not required more than 2 changes in their ART regimen.
* ALT or aspartate aminotransferase (AST) values >1.5 x ULN during Screening/Baseline.
* Total bilirubin values >1.0 x ULN during Screening/Baseline.
* History of drug or alcohol abuse in the 2 years prior to Screening.
* Any malignancy within the 5 years prior to Screening except for basal cell carcinoma successfully treated with local therapy.
* Medical history or findings that preclude safe participation in the study or who are likely to be non-compliant with study procedures in the opinion of the Investigator or medical monitor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Chapman, MD, Principal Investigator — University of Chicago, Chicago, IL USA
Locations (6):
- United States (6):
  - University of California Los Angeles, Los Angeles, California
  - University of Chicago Medicine & Biological Sciences, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - Nephrology Associates of Northern Virginia, Inc., Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fontana RJ, Watkins PB, Bonkovsky HL, Chalasani N, Davern T, Serrano J, Rochon J; DILIN Study Group. Drug-Induced Liver Injury Network (DILIN) prospective study: rationale, design and conduct. Drug Saf. 2009;32(1):55-68. doi: 10.2165/00002018-200932010-00005. PMID 19132805

RESULTS

PARTICIPANT FLOW:
Groups:
- Lixivaptan: After meeting entry criteria during a 1-3-week Screening Period, participants entered a 3-week no study drug Baseline Period to obtain baseline measurements.
  All participants who completed the Pre-Titration period entered a 3-6 week Titration Period following the Baseline Period, during which each individual participant was titrated with oral lixivaptan capsules administered twice daily to a dose that was tolerated and resulted in a reduced trough urine specific gravity (or until the maximum dose level was reached) for each individual. The minimum dose to enter the Maintenance Period was 100 mg BID, and the maximum was 200 mg BID. Treatment in the Maintenance Period was continued for up to 52 weeks.
Period: Baseline Period (No Treatment)
Arm/Group | Lixivaptan
Started | 7
Completed | 6
Not Completed | 1
Not completed — Baseline Failure | 1
Period: Titration Period
Arm/Group | Lixivaptan
Started | 6
Completed | 6
Not Completed | 0
Period: Maintenance Period
Arm/Group | Lixivaptan
Started | 6
Completed | 2
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Sponsor Termination of Study | 2
Period: Follow-up Period
Arm/Group | Lixivaptan
Started | 6 (All participants who were treated with Lixivaptan completed the Follow-up Period, including those who did not complete the Maintenance Period.)
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: Baseline data were obtained from the Safety Population, which consisted of all participants who were treated with lixivaptan.
Arm/Group | Safety Population
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.70 (3.107)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Develop Serum Alanine Aminotransferase (ALT) Levels >3 × ULN During the Titration or Maintenance Periods Assessed to be Related to Lixivaptan and Result in Discontinuation of Lixivaptan Treatment
Description: Number of participants who develop serum ALT levels >3 x ULN which are assessed by the independent Hepatic Events Review Committee (HERC) to be at least probably related to lixivaptan and result in the discontinuation of lixivaptan treatment. The independent HERC, after reviewing demographic, medical and medication history, safety data and other relevant data of participants who develop liver abnormalities, will determine the probable causality for liver chemistry test abnormalities of concern and the relatedness to lixivaptan using the Drug-Induced Liver Injury Network probability criteria (Fontana et al., 2009). The normal range of ALT was defined as 0-55 U/L.
Time Frame: Up to 58 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Lixivaptan: Titration and Maintenance Periods: All participants who successfully completed the Baseline Period entered a 3-6-week Titration Period, during which each individual participant was titrated with oral lixivaptan capsules administered twice daily to a dose that was tolerated and resulted in a reduced trough urine specific gravity (or until the maximum dose level was reached) for each individual. The minimum dose to enter the Maintenance Period was 100 mg BID, and the maximum was 200 mg BID. Treatment in the Maintenance Period was continued for up to 52 weeks.
Arm/Group | Lixivaptan: Titration and Maintenance Periods
Number analyzed (Participants) | 6
Participants | 1

2. Secondary Outcome: Number of Participants Who Develop Serum ALT Levels >5 × ULN During the Titration or Maintenance Periods Assessed to be Related to Lixivaptan and Result in Discontinuation of Lixivaptan Treatment
Description: Number of participants who develop serum ALT levels >5 x ULN which are assessed by the independent HERC to be at least probably related to lixivaptan and result in the discontinuation of lixivaptan treatment. The independent HERC, after reviewing demographic, medical and medication history, safety data and other relevant data of participants who develop liver abnormalities, will determine the probable causality for liver chemistry test abnormalities of concern and the relatedness to lixivaptan using the Drug-Induced Liver Injury Network probability criteria (Fontana et al., 2009). The normal range of ALT was defined as 0-55 U/L.
Time Frame: Up to 58 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lixivaptan: Titration and Maintenance Periods
Number analyzed (Participants) | 6
Participants | 1

3. Secondary Outcome: Number of Participants Who Develop Serum ALT Levels >3 × ULN During the Titration or Maintenance Periods Assessed to be Related to Lixivaptan and Result in Dose Reduction of Lixivaptan Treatment
Description: Number of participants who develop serum ALT levels >3 x ULN which are assessed by the independent HERC to be at least probably related to lixivaptan and result in the dose reduction of lixivaptan treatment. The independent HERC, after reviewing demographic, medical and medication history, safety data and other relevant data of participants who develop liver abnormalities, will determine the probable causality for liver chemistry test abnormalities of concern and the relatedness to lixivaptan using the Drug-Induced Liver Injury Network probability criteria (Fontana et al., 2009). The normal range of ALT was defined as 0-55 U/L.
Time Frame: Up to 58 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lixivaptan: Titration and Maintenance Periods
Number analyzed (Participants) | 6
Participants | 0

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs during the Titration Period, the Maintenance Period, or the Follow-up Period.
Time Frame: Up to 62 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Lixivaptan: Titration, Maintenance, and Follow-up Periods: Participants in this group are those who completed the Titration Period, entered the Maintenance Period (regardless of whether they completed it), and completed the Follow-up Period.
Arm/Group | Lixivaptan: Titration, Maintenance, and Follow-up Periods
Number analyzed (Participants) | 6
Participants
  Titration and Maintenance Periods | 6
  Follow-up Period | 1

5. Secondary Outcome: Number of Participants With Potentially Clinically Important Clinical Laboratory Findings
Description: Number of participants with clinical laboratory findings (non-hepatic clinical chemistry, hematology, and urinalysis) recorded during the Titration Period, the Maintenance Period, or the Follow-up Period, and considered to be potentially clinically important.
Time Frame: Up to 62 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lixivaptan: Titration, Maintenance, and Follow-up Periods
Number analyzed (Participants) | 6
Participants
  Titration and Maintenance Periods | 1
  Follow-up Period | 0

6. Secondary Outcome: Number of Participants With Potentially Clinically Important Vital Signs Findings
Description: Number of participants with vital signs findings (heart rate, diastolic and systolic blood pressure, weight) recorded during the Titration Period, the Maintenance Period, or the Follow-up Period, and considered to be potentially clinically important.
Time Frame: Up to 62 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lixivaptan: Titration, Maintenance, and Follow-up Periods
Number analyzed (Participants) | 6
Participants
  Titration and Maintenance Periods | 5
  Follow-up Period | 0

7. Secondary Outcome: Number of Participants With Potentially Clinically Important 12-lead Electrocardiogram (ECG) Findings
Description: Number of participants with ECG findings recorded during the Titration Period, the Maintenance Period, or the Follow-up Period, and considered to be potentially clinically important (defined as a QT interval corrected for heart rate according to Fridericia's formula [QTcF] ≥ 450 msec).
Time Frame: Up to 62 weeks
Population: The same participant experienced potentially clinically important ECG findings in the Baseline Period, in addition to during the Titration and Maintenance, and Follow-up Periods.
Measure: Count of Participants; unit: Participants
Arm/Group | Lixivaptan: Titration, Maintenance, and Follow-up Periods
Number analyzed (Participants) | 6
Participants
  Baseline Period | 1
  Titration and Maintenance Periods | 1
  Follow-up Period | 1

8. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR) From Baseline to Final Assessment
Description: Baseline eGFR is defined as the mean of the 3 eGFR assessments obtained during the Baseline Period (if any values are missing, the remaining values will be used to determine the baseline eGFR). The endpoint eGFR is defined as the mean of 3 eGFR assessments obtained during the Follow-up Period (if any values are missing, the remaining values will be used to determine the endpoint eGFR). The change in eGFR from Baseline to Final Assessment will be provided.
Time Frame: Up to 62 weeks
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Lixivaptan: Titration, Maintenance, and Follow-up Periods
Number analyzed (Participants) | 6
mL/min/1.73m^2 | -4.3 (2.7)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from when participants had taken their first dose of lixivaptan in the Titration Period until the end of the study (maximum duration: 455 days)
Groups:
- Titration and Maintenance Periods: All participants who completed the Titration Period and entered the Maintenance Period
- Follow-up Period: All participants who entered the Follow-up Period, regardless of whether they had completed the Maintenance Period
Arm/Group | Titration and Maintenance Periods | Follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Titration and Maintenance Periods (N=6) | Follow-up Period (N=6)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Titration and Maintenance Periods (N=6) | Follow-up Period (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Efficacy and safety results are limited by the early termination of the trial and the small number of subjects. Early termination was due to a sponsor decision for reasons unrelated to safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT04152837/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT04152837/SAP_001.pdf